CLINICAL TRIAL: NCT00151216
Title: Administration of a Replication Deficient Adeno-associated Virus Gene Transfer Vector Expressing the Human CLN2 cDNA to the Brain of Children With Late Infantile Neuronal Ceroid Lipofuscinosis
Brief Title: Safety Study of a Gene Transfer Vector for Children With Late Infantile Neuronal Ceroid Lipofuscinosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Nathan's Battle Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0401007010; OBA-RAC 0312-619 (Other: Office of Biotechnology Activities - Recombinant DNA)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Batten Disease; Late Infantile Neuronal Ceroid Lipofuscinosis
Keywords: Batten Disease; Late Infantile Neuronal Ceroid Lipofuscinosis; LINCL
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Intervention Model Description: The study will be carried out in two populations of children with LINCL. Group A will include n= 5 children with a total disability score of 0 to 4 (the severe forms of the disease; the staging based on a modification of the scale of Steinfeld et al. Group B will include n=6 children with a total disability score of 5 to 6, a moderate stage of the disease. All of the study population of 11 children (Group A, n= 5 and Group B, n=6) will receive 3x10^12 particle units of the AAV2CUhCLN2 vector divided among 12 locations delivered through 6 burr holes (2 locations at varying depths through each hole), 3 burr holes per hemisphere. The choice of the locations for the burr holes and needle placement will be on a case-by-case basis due to the diffuse and variable nature of the disease presentation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A-Severe Stages of LINCL (Experimental): Group A will include n= 5 children with a total disability score of 0 to 4 (the severe forms of the disease; the staging based on a modification of the scale of Steinfeld et al.
  All subjects will receive 3x10^12 particle units of the AAV2CUhCLN2 vector.
  Interventions: Biological: AAV2CUhCLN2 (3x10^12 particle units)
- Group B-Moderate Stages of LINCL (Experimental): Group B will include n=6 children with a total disability score of 5 to 6, a moderate stage of the disease.
  All subjects will receive 3x10^12 particle units of the AAV2CUhCLN2 vector.
  Interventions: Biological: AAV2CUhCLN2 (3x10^12 particle units)

INTERVENTIONS:
Biological: AAV2CUhCLN2 (3x10^12 particle units) — gene transfer; one-time administration via neuro surgery procedure

SUMMARY:
The aim of this study is to treat the signs and symptoms of late infantile neuronal ceroid lipofuscinosis (LINCL), a fatal inherited disease in the brain. This will be accomplished by using delivery of a gene (method called gene transfer) to administer to the brain an experimental drug called AAV2CUhCLN2, a gene transfer vector.

DETAILED DESCRIPTION:
Late infantile neuronal ceroid lipofuscinosis (LINCL) is a fatal childhood neurodegenerative lysosomal storage disease with no known therapy. There are estimated to be 200 to 300 children in the USA at any one time with the disease. LINCL is a genetic disease resulting from mutations in the CLN2 gene. The CLN2 gene encodes a protein tripeptidyl peptidase-I (TPP-I) which is absent/deficient in children with LINCL. This absence/deficiency of TPP-I results in lysosomal storage and subsequent cell death (especially neurons). The children with LINCL are chronically ill, with a progressive CNS disorder that invariably results in death, typically by age 8 to 12.

This clinical study will evaluate the concept that persistent expression of the normal CLN2 cDNA in the CNS will result in the production of sufficient amounts of TPP-I to prevent further loss of neurons, and hence limit disease progression. To assess this concept, an adeno-associated virus vector encoding the normal human CLN2 gene (AAV2CUhCLN2) will be used as a vehicle to deliver and express the human CLN2 cDNA in the brain of children with LINCL. The proposed study will include 11 individuals and will be divided into two parts. Group A, to be studied first, will include 5 individuals with the severe form of the disease. Group B of the trial will include 6 individuals with a moderate form of the disease. Following direct intracranial administration of the vector, there will be neurological assessment using the LINCL clinical rating scale and magnetic resonance imaging/magnetic resonance spectroscopy assessment of the CNS in regions of vector administration. The data generated will help evaluate two hypotheses: (1) that it is safe to carry out direct intracranial administration of the AAV2CUhCLN2 vector to the CNS of individuals with LINCL; and (2) that administration of the AAV2CUhCLN2 vector will slow down or halt the progression of the disease in the central nervous system.

ELIGIBILITY:
Inclusion Criteria:

* A definitive diagnosis of late infantile neuronal ceroid lipofuscinosis, based on clinical phenotype and genotype, with CLN2 gene mutations known to be associated with the disease.
* All subjects will be naive, i.e., they have not previously participated in a gene therapy study for LINCL.
* Parents of study participants must agree to comply in good faith with the conditions of the study, including attending all of the required baseline and follow-up assessments.
* Both parents or legal guardians must give consent for their child's participation in the research study.
* For group A, subjects will have a LINCL average total disability score 0 to 4, the severe form of the disease.
* For group B, subjects will have a LINCL average total disability score 5 to 6, a moderate form of the disease.

Exclusion criteria

* Other significant medical or neurological conditions may disqualify the patient from participation in this study, particularly those which would create an unacceptable operative risk or risk to receiving the AAV2CUhCLN2 vector. Examples include malignancy (other than skin cancer), congenital heart disease, liver or renal failure, or seropositive for HIV. Each case will be individually reviewed and the final decision shall rest with the Eligibility Committee comprised on three physicians other than the Principal Investigator, including a pediatric neurosurgeon, pediatric neurologist and general pediatrician.
* Individuals without adequate control of seizures (i.e., a seizure score <3 on the CNS Disability Scoring System for Late Infantile Neuronal Ceroid Lipofuscinosis).
* Individuals with heart disease that would be a risk for anesthesia.
* History of hemorrhage or major risk factors for hemorrhage (e.g., abnormally low platelet counts).
* Concurrent participation in any other FDA approved Investigational New Drug clinical protocol is not allowed, although the Principal Investigator will work with other doctors to accommodate specific requests (e.g., a study of nutritional supplements probably would not be a disqualification).
* Individuals who have a (1) heart pacemaker and/or related implants, (2) metal fragment/chip in the eye or other sites, (3) an aneurysm clip in their brain, and (4) metallic inner ear implants.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2004-06; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Neurological assessment using the LINCL clinical rating scale | screening; pre-therapy; and 6 and 18 months post-vector administration
  The neurological examination will be carried out using a standard format with input from the parents/legal guardians as relevant. The clinical rating scale, referred to as a "CNS disability scale" is made up of individual sum of 4 point scales for each of 3 activities; the ratings for each activity are summed, giving a "CNS disability score". Each of the activities are rated 0 to 3, where 0 is the most severe form of the disease. This scale, developed by Steinfeld et al, originally included the four major functional problems in LINCL (loss of motor performance, seizure activity, loss of vision, and loss of language). In this modified clinical rating system, these are now 3 categories.

SECONDARY OUTCOMES:
MRI/MRS assessment | screening; pre-therapy; and 6 and 18 months post-vector administration
  The secondary endpoint variable will be the MRI/MRS assessment of the CNS in regions of vector administration. Anatomical measurements of brain parenchymal volume will be combined with proton spectroscopic imaging of the n-acetyl-aspartate (NAA) resonance, a neuronal marker measurable using clinical magnetic resonance techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G. Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital - Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sondhi D, Kaminsky SM, Rosenberg JB, Rostami MR, Hackett NR, Crystal RG. Twenty-Year Survival Analysis of Adeno-Associated Virus Vector Serotype 2-Mediated Gene Therapy to the Central Nervous System for CLN2 Disease. Hum Gene Ther. 2024 Jan;36(1-2):28-35. doi: 10.1089/hum.2024.182. Epub 2025 Jan 2. PMID 39745261
- [Derived] Worgall S, Sondhi D, Hackett NR, Kosofsky B, Kekatpure MV, Neyzi N, Dyke JP, Ballon D, Heier L, Greenwald BM, Christos P, Mazumdar M, Souweidane MM, Kaplitt MG, Crystal RG. Treatment of late infantile neuronal ceroid lipofuscinosis by CNS administration of a serotype 2 adeno-associated virus expressing CLN2 cDNA. Hum Gene Ther. 2008 May;19(5):463-74. doi: 10.1089/hum.2008.022. PMID 18473686